CLINICAL TRIAL: NCT00195104
Title: Phase I/II Study of Arsenic Trioxide in Combination With Cytosine Arabinoside in Patients With High-risk Myelodysplastic Syndrome and Poor-prognosis Acute Myelogenous Leukemia
Brief Title: Arsenic Trioxide in Combination With Cytarabine in Patients With High-risk MDS and Poor-prognosis AML
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0603-887
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Arsenic Trioxide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Patients (Experimental): Arsenic trioxide [TrisenoxTM Injection], 0.25mg/kg/dose administered intravenously over 1 to 4 hours
  Interventions: Drug: Arsenic Trioxide (Tricenox); Drug: Cytarabine

INTERVENTIONS:
Drug: Arsenic Trioxide (Tricenox)
Drug: Cytarabine

SUMMARY:
The purpose of this study is to find out the effectiveness and side effects of arsenic trioxide in combination with low-dose ara-C.

DETAILED DESCRIPTION:
This is an open-label, single institution, dose-escalation study of low-dose cytosine arabinoside and arsenic trioxide.

Patients will receive a fixed dose of arsenic trioxide administered 0.25mg/kg/day on days 1-5 and 8-12 and ara-C administered at 5, 7.5, or 10 mg/m2 SC BID days 1-14 in repeated cycles of 2 weeks on therapy and 2 weeks off therapy in a standard dose escalation design (1 cycle = 2 weeks on therapy + 2 weeks off therapy).

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of high-risk MDS (IPSS int-2).
* No prior cytotoxic therapy for MDS or AML (patients may have received prior therapy with hematopoietic growth factors, immunomodulatory agents or 5-azacitidine).

Exclusion Criteria:

* Pregnant or lactating women.
* Absolute QT interval >460 msec in the presence of serum potassium and magnesium values within the normal range.
* Concurrent treatment with maintenance therapy, cytotoxic chemotherapy, radiation, or investigational agents.
* Uncontrolled or severe cardiovascular or pulmonary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2003-09-17 (Actual); Primary Completion 2006-03-17 (Actual); Study Completion 2006-06-20 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of cytosine arabinoside in combination with ATO 0.25mg/kg/day IV for 10 days on therapy followed by 14 days off therapy in patients with high-risk MDS and poor-prognosis AML. | 10 days on therapy followed by 14 days off therapy in patients with high-risk MDS and poor-prognosis AML
To characterize the safety and tolerability of the combination of ATO and low-dose ara-C, including acute and chronic toxicities. | 4 weeks after the last study treatment

SECONDARY OUTCOMES:
To determine the CR and PR rates in patients with high-risk MDS and poor-prognosis AML treated with the combination of ATO and low-dose ara-C. | 4 weeks after the last study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gail Roboz, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medcial College of Cornell University, New York, New York, United States

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/20956016